CLINICAL TRIAL: NCT00907751
Title: Association of Rituximab to Plasma Exchange in Adult Acquired Idiopathic Thrombotic Thrombocytopenic Purpura
Brief Title: Rituximab in Adult Acquired Idiopathic Thrombotic Thrombocytopenic Purpura
Acronym: PTTritux
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060801
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Microangiopathic hemolytic anemia (< 12 g/dL) with thrombocytopenia (<50 G/L)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — Patients will be treated according to the recommendations of the Reference Centre for the management of thrombotic microangiopathies. Infusions of rituximab (375 mg/m2) will be added to this treatment at day 1, 4 and 15, immediately after plasma exchange sessions.

SUMMARY:
Multicentric non-randomized phase II opened prospective study (10 centres involved).

Primary endpoint:

* To evaluate the kinetics of B-cell depletion by rituximab and its pharmacokinetics in patients treated with rituximab in association with plasma exchanges.

Secondary endpoints:

* To evaluate the tolerance of rituximab, the volume of plasma and the number of plasma exchange sessions required to achieve a durable complete remission, and to determinate the duration of B-cell depletion.
* To evaluate the incidence of persistent severe acquired ADAMTS13 deficiency following treatment with rituximab, as well as the incidence of relapses.

DETAILED DESCRIPTION:
Duration of the study:

3 years and 2 months, including 1 year of inclusion and 2 years of participation for the patient.

Experimental plan:

Patients fulfilling the inclusion criteria of the study will be treated according to the recommendations of the Reference Centre for the management of thrombotic microangiopathies. If patients present refractory TTP, infusions of rituximab (375 mg/m2) will be added to this treatment at day 1, 4 and 15, immediately after plasma exchange sessions.On diagnosis, during treatment and after remission achievement, the following values will be explored: ADAMTS13 activity, ADAMTS13 inhibitors and anti-ADAMTS13 antibodies, B-cell lymphocytes quantification by immunophenotyping, and serum gammaglobulin level by serum protein electrophoresis. Rituximab will also be quantified.

Number of patients:

Each participating centre may recruit and include 1 patient/year.Amongst 10 participating centres, a total number of 10 patients should be included.

Specific activities during the study:

Three infusions of rituximab (375 mg/m2 /infusion), immediately after plasma exchange sessions on day 1, 4 and 15. Blood samplings at day 1, 4 and 15, at 1 month and then every 3 month until month 24.

Expected results and perspectives:

This study should provide evidence as to whether the association of rituximab to plasma exchanges allo an efficient B-cell depletion. If yes, a randomized study should be performed to evaluate the role of rituximab at the acute phase of acquired idiopathic TTP, immediately after the diagnosis was established.

ELIGIBILITY:
Inclusion Criteria:

* Microangiopathic hemolytic anemia (< 12 g/dL) with thrombocytopenia <50 G/L, and mild or no renal failure (Serum creatinine < 150 µmol/L),
* negative Beta HCG and ongoing contraception during treatment and during the 24 months following the last infusion of rituximab,
* refractory TTP (after 4 days of standard treatment)
* > 18 year old
* and signed written informed consent.

Exclusion Criteria:

* Hemolytic uremic syndrome (platelet count ³ 50 G/L and serum creatinine ³ 150 micromol/L),
* TTP associated with another condition (HIV infection, cancer and/or chemotherapy, transplantation),
* previous treatment with vincristine or cyclophosphamide or other immunomodulatory drugs (except steroids), within 2 months before inclusion ;
* ongoing or planned pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the kinetics of B-cell depletion by rituximab and its pharmacokinetics in patients treated with rituximab in association with plasma exchanges | at 1, 3, 6, 9, 12, 18 and 24 months

SECONDARY OUTCOMES:
To evaluate the tolerance of rituximab, the volume of plasma and the number of plasma exchange sessions required to achieve a durable complete remission, and to determinate the duration of B-cell depletion | at 1, 3, 6, 9, 12, 18 and 24 months
To evaluate the incidence of persistent severe acquired ADAMTS13 deficiency following treatment with rituximab, as well as the incidence of relapses. | at 1, 3, 6, 9, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul COPPO, Md Ph D, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Saint-Antoine Hospital, Hematology, Paris, France

REFERENCES:
- [Derived] Benhamou Y, Paintaud G, Azoulay E, Poullin P, Galicier L, Desvignes C, Baudel JL, Peltier J, Mira JP, Pene F, Presne C, Saheb S, Deligny C, Rousseau A, Feger F, Veyradier A, Coppo P; French Reference Center for Thrombotic Microangiopathies. Efficacy of a rituximab regimen based on B cell depletion in thrombotic thrombocytopenic purpura with suboptimal response to standard treatment: Results of a phase II, multicenter noncomparative study. Am J Hematol. 2016 Dec;91(12):1246-1251. doi: 10.1002/ajh.24559. Epub 2016 Nov 8. PMID 27643485